CLINICAL TRIAL: NCT06219005
Title: Standardized Assessment of Emergency Physician Ultrasound-guided Nerve Block Training Using a Low-fidelity Simulation Model
Brief Title: Ultrasound-guided Nerve Block Training Model and Evaluation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00114989
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-04

CONDITIONS: Nerve Blocks; Medical Education, Simulation, Crisis Resource Management; Medical Education in Emergency Ultrasound

STUDY DESIGN:
Intervention Model Description: prospective observational cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency Medicine attending physicians and residents (Experimental)
  Interventions: Behavioral: ultrasound education and simulation workshop

INTERVENTIONS:
Behavioral: ultrasound education and simulation workshop — workshop testing emergency physician knowledge and technical skills in performing ultrasound-guided nerve blocks in a simulation model

SUMMARY:
The aim of this study is to assess emergency medicine physician knowledge and technical skill in performance of ultrasound-guided serratus anterior nerve block in a low-fidelity simulation model workshop and to determine the feasibility, acceptability, and usability of the training program. By performing this study, the investigators hope to create a standardized training model which could potentially facilitate POCUS and critical procedural performance and thereby improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine attending and resident physicians

Exclusion Criteria:

* ED nursing, ED technicians, and advanced practice physicians (APPs)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Physician knowledge assessment | 4 months
  The investigators will assess ultrasound-guided serratus anterior nerve block in a simulation model using surveys at 1 month pre-intervention, post-intervention, and 3 months post-intervention (Likert scale 0-5 with values of Strongly disagree, disagree, neutral, agree, strongly agree)
Physician technical skills assessment | 4 months
  The investigators will assess ultrasound-guided serratus anterior nerve block in a simulation model using surveys at 1 month pre-intervention, post-intervention, and 3 months post-intervention (Likert scale 0-5 with values of Strongly disagree, disagree, neutral, agree, strongly agree).

SECONDARY OUTCOMES:
acceptability of our implementation strategy | 4 months
  The investigators will evaluate EM physician education and simulation workshop implementation strategy acceptability using a post-intervention survey (Likert scale 0-5 with values of Strongly disagree, disagree, neutral, agree, strongly agree).
appropriateness of our implementation strategy | 4 months
  The investigators will evaluate EM physician education and simulation workshop implementation strategy appropriateness using a post-intervention survey (Likert scale 0-5 with values of Strongly disagree, disagree, neutral, agree, strongly agree).
feasibility of our implementation strategy | 4 months
  The investigators will evaluate EM physician education and simulation workshop implementation strategy feasibility using a post-intervention survey (Likert scale 0-5 with values of Strongly disagree, disagree, neutral, agree, strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
All participant information will be confidential and restricted to the research study team. Deidentified summary data will be made available after study completion for public and scientific community dissemination and future clinical improvements.

REFERENCES:
- [Background] Petrosoniak A, Herold J, Woolfrey K. Emergency medicine procedural skills: what are residents missing? CJEM. 2013 Jul;15(4):241-8. doi: 10.2310/8000.2013.130897. PMID 23777999
- [Background] Sherbino J, Bandiera G, Frank JR. Assessing competence in emergency medicine trainees: an overview of effective methodologies. CJEM. 2008 Jul;10(4):365-71. doi: 10.1017/s1481803500010381. PMID 18652729
- See also: ACEP emergency ultrasound guidelines — https://www.acep.org/patient-care/policy-statements/ultrasound-guidelines-emergency-point-of--care-and-clinical-ultrasound-guidelines-in-medicine
- See also: IFEM point-of-care-ultrasound guidelines — https://www.ifem.cc/point_of_care_ultrasound_curriculum_guidelines